CLINICAL TRIAL: NCT00674180
Title: Data Analysis of a Managed Care Weight Reduction Trial
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Judith Wylie-Rosett, Prof. Epidemiology & Population Health, Albert Einstein College of Medicine
Other Study IDs: 2008-833
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: a workbook alone
  Interventions: Behavioral: Workbook
- 2: a workbook alone and the addition of computerized tailoring using onsite computer kiosks with touch screen monitors
  Interventions: Behavioral: Workbook; Behavioral: Computer Intervention
- 3: a workbook, the addition of computerized tailoring using onsite computer kiosks with touch screen monitors, and staff consultations.
  Interventions: Behavioral: Workbook; Behavioral: Computer Intervention; Behavioral: Staff Consultation

INTERVENTIONS:
Behavioral: Workbook — The workbook developed as a do-it-yourself program in which participants completed self-help sheets that guided them to sections of the workbook most salient to their needs.
Behavioral: Computer Intervention — The computer intervention was provided using a network system that included a file server plus 5 multimedia computers with touch screens. The expert software program was written to guide participants in using the workbook and tail behavioral goals based on their prior computer use and the answers they provided on baseline questionnaires. The three primary paths in the computer addressed nutrition, fitness, and psychobehavioral content.
  Groups: 2; 3
Behavioral: Staff Consultation — The staff consultation component included 6 closed-group workshop sessions and up to 18 telephone or face-to-face consultations with a registered dietician and/or a cognitive behavioral therapist. The workshop curriculum focused on specific activities and assignments in the workbook, and it encouraged use of the computer to identify problems and issues.
  Groups: 3

SUMMARY:
This study will involve secondary data analysis for a study done by Wylie-Rosett et al. in 2001 that evaluated the costs and effects of incremental components of a weight-loss program. Data analysis will involve cross-sectional and predictive analyses and may include: regression analyses to determine predictors of weight loss and cardiovascular risk, correlations between weight reduction strategies and biological indices, and interactions between biomarkers of inflammation and traditional cardiovascular risk factors. This data will also be available for economic modeling.

DETAILED DESCRIPTION:
This study will involve secondary data analysis for a study done by Wylie-Rosett et al. in 2001. Using a 3-arm, 12-month randomized clinical trial, Wylie-Rosett et al. evaluated the costs and effects of incremental components of a weight-loss program. The study included 588 individuals (BMI> 25 kg/m2) in a freestanding health maintenance organization and achieved an 81% completion rate. The intervention used a cognitive behavioral approach for tailoring lifestyle modification goals. The incremental levels of interventions included a) a workbook alone, b) the addition of computerized tailoring using onsite computer kiosks with touch screen monitors, and c) the addition of both computers and staff consultations. For the increasing levels of intervention intensity, the mean 12-month weight losses were 2.2, 4.7, and 7.4 pounds, with the respective cost per participant being $12.33, $41.99, and $133.74. The decreases in mean BMIs for these respective intervention levels were 0.4, 0.9, and 1.2. All groups reported a decrease in energy and fat intake and an increase in blocks walked (p<.01). Intervention variables that correlated with weight loss included more computer logons, achieving computer-selected goals, more self-monitoring, increased walking, and decreased energy and fat intake, as well as higher attendance in staff consultation group sessions for that treatment condition. Weight loss correlated with decreases in fasting glucose and blood pressure. Wylie-Rosett et al. (2001) concluded that, in a weight-loss program, computers can facilitate selecting behavioral change goals. More frequent usage resulted in greater weight loss, and staff counseling to augment the computer intervention achieved the most weight loss. The purpose of this study will be secondary analysis of the data collected in the original MODELS study.

ELIGIBILITY:
Inclusion Criteria:

* BMI of more than 25 (or a BMI of 24 or more plus 1 cardiovascular risk factor), and the willingness to follow the study protocol, which included a refundable $100 deposit

Exclusion Criteria:

* Intention to move beyond commuting distance in the next 12 months,
* Medical conditions that would interfere with study participation,
* Unwillingness to follow the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants were recruited from an HMO's patient population and from New Hyde Park, NY.
Sampling Method: Non-Probability Sample
Enrollment: 588 (Actual)
Dates: Start 2008-04; Primary Completion 2008-04 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
weight loss | 1 year

SECONDARY OUTCOMES:
diabetes and cardiovascular risk | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Judith Wylie-Rosett, EdD, Principal Investigator — Albert Einstein College of Medicine; Charles Swencionis, PhD, Study Chair — Yeshiva University

REFERENCES:
- [Result] Wylie-Rosett J, Swencionis C, Ginsberg M, Cimino C, Wassertheil-Smoller S, Caban A, Segal-Isaacson CJ, Martin T, Lewis J. Computerized weight loss intervention optimizes staff time: the clinical and cost results of a controlled clinical trial conducted in a managed care setting. J Am Diet Assoc. 2001 Oct;101(10):1155-62; quiz 1163-4. doi: 10.1016/s0002-8223(01)00284-x. PMID 11678486
- [Derived] Swencionis C, Wylie-Rosett J, Lent MR, Ginsberg M, Cimino C, Wassertheil-Smoller S, Caban A, Segal-Isaacson CJ. Weight change, psychological well-being, and vitality in adults participating in a cognitive-behavioral weight loss program. Health Psychol. 2013 Apr;32(4):439-46. doi: 10.1037/a0029186. Epub 2012 Aug 13. PMID 22888821